CLINICAL TRIAL: NCT01458795
Title: The Fate Of Calf Perforators After Endovenous Laser Ablation Of Saphenous Veins
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ugur Ozkan, MD, Associate professor of radiology, Baskent University
Allocation: Non-Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: bask 012
Record Dates: First submitted 2011-10-20; First posted 2011-10-25 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Endovenous laser ablation

SUMMARY:
The aim of this study is to evaluate the morphologic and hemodynamic changes in the calf perforators after endovenous laser ablation of saphenous veins.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients who undergo EVLA procedure for saphenous vein insufficiency

Exclusion Criteria:

* Patients with a history of deep venous thrombosis (DVT)
* Previous varicose vein surgery or injection sclerotherapy
* Patients without superficial venous incompetency

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Adana, Turkey (Türkiye)